CLINICAL TRIAL: NCT03501680
Title: Randomized, Controlled, Open-label Trial of Intravenous Intensive Insulin for Severe/Moderate Hypertriglyceridemia Pancreatitis.
Brief Title: Intensive Insulin for Severe/Moderate Hypertriglyceridemia Pancreatitis.
Acronym: HAPinsulin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Meng-Tao Zhou, The director of the department of pancreatitis; the president of First Affiliated Hospital of Wenzhou Medical Univeristy, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAPinsulin
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Acute Pancreatitis; Hypertriglyceridemia
Keywords: hyperlipidaemic pancreatitis; Plasmapheresis; insulin
MeSH Terms: conditions — Pancreatitis; Hypertriglyceridemia; Insulin Resistance | interventions — Insulin; Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Group A: intensive insulin (Experimental): Group A: intensive insulin (glycemic control 4.4-6.1mmol/L)
  Interventions: Drug: Insulin
- Group B: standard insulin (Active Comparator): Group B: standard insulin (glycemic control 7.8-10.0 mmol/L),
  Interventions: Drug: Insulin
- Group C: plasmapheresis (Active Comparator): Group C: plasmapheresis
  Interventions: Device: plasmapheresis

INTERVENTIONS:
Drug: Insulin — Group A: intensive insulin (glycemic control 4.4-6.1mmol/L), Group B: standard insulin (glycemic control 7.8-10.0 mmol/L), and Group C: plasmapheresis.
  Insulin was injected by insulin pump.
  Arms: Group A: intensive insulin; Group B: standard insulin
Device: plasmapheresis — Triglyceridemia should be less than 5.65 mmol/l.
  Arms: Group C: plasmapheresis

SUMMARY:
The aim of this study is to investigate the therapeutic efficacy of intensive insulin in patients with hypertriglyceridemia induced moderate/severe acute pancreatitis on the course and outcome of disease.

DETAILED DESCRIPTION:
Hypertriglyceridemia-induced acute pancreatitis occurs in about 1-4% of the cases. It is the third leading cause of pancreatitis after biliary and alcoholic etiology. Hypertriglyceridemia can be caused by primary causes, lipid metabolism disorders and secondary causes.

Hyperlipidemic pancreatitis can be provoked when triglyceride levels (TGL) exceed 11.3 mmol/l (1,000 mg/dl). Except for standard symptomatic treatment, plasmapheresis and insulin have been performed to rapidly reduce TGL and chylomicron levels in the blood.The therapeutic efficacy of intensive insulin, standard insulin, and plasmapheresis in patients with hypertriglyceridemia induced moderate/severe acute pancreatitis on the course and outcome of disease.After acceptance patients will be randomized by random envelope in the 3 groups: Group A: intensive insulin (glycemic control 4.4-6.1mmol/L), Group B: standard insulin (glycemic control 7.8-10.0 mmol/L), and Group C: plasmapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertriglyceridemia induced acute pancreatitis (AP): Typical pain increase in serum lipase or amylase with serum TG> 1,000 mg/dL (11.3mmol/L) or serum was milky with serum TG> 500 mg/dL(5.65 mmol/L)
* Onset of abdominal pain within <=48h before admission
* moderate severe or severe Acute Pancreatitis according to Atlanta criteria
* except for other AP causes, such as cholelithiasis, alcohol, drugs and so on

Exclusion Criteria:

* other etiologies other than hyperlipidemia leading to AP
* at the same time combined with other etiologies of AP
* appear difficult to reverse respiratory failure, severe systemic circulatory failure, coma and other the endangered symptoms, patients expected to die within 24hours
* disseminated intravascular coagulation, or patients with severe active bleeding
* without informed consent, the patient refused to plasma replacement, and other circumstances may bring significant bias.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-06 (Estimated); Primary Completion 2020-03-08 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of mortality | From admition to hospital discharge, an average of 2 months
  Number of participants with fatal outcome during hospitalisation
Reduction of organ failure | From admition to hospital discharge, an average of 2 months
  reanl failure, respiratory failure, circulatory failure etal
triglyceride levels | From admition to hospital discharge, an average of 2 months
  triglyceride levels

SECONDARY OUTCOMES:
cytokines in serum, urine | From admition to 7 days
  IL-6, IL-8, IL-10
insulin dose | From admition to 7 days
  insulin dose
Severity Score in CT scan | From admition to 7 days
  CT Balthazar score/grade or MCTSI score
TNF-α in serum, urine | From admition to 7 days
  TNF-α
Clinical Severity Score | From admition to 7 days
  BISAP score

OTHER OUTCOMES:
Genomics | From admition to 7 days
  cfDNA et.al.
Clinical Severity Score | From admition to 7 days
  Ranson score
Clinical Severity Score | From admition to 7 days
  Apache2

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Tao Zhou, M.D., Study Director — The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lutfi R, Huang J, Wong HR. Plasmapheresis to treat hypertriglyceridemia in a child with diabetic ketoacidosis and pancreatitis. Pediatrics. 2012 Jan;129(1):e195-8. doi: 10.1542/peds.2011-0217. Epub 2011 Dec 26. PMID 22201145
- [Background] Tsuang W, Navaneethan U, Ruiz L, Palascak JB, Gelrud A. Hypertriglyceridemic pancreatitis: presentation and management. Am J Gastroenterol. 2009 Apr;104(4):984-91. doi: 10.1038/ajg.2009.27. Epub 2009 Mar 17. PMID 19293788